CLINICAL TRIAL: NCT02451215
Title: LITT for the Treatment of Newly Diagnosed Central Nervous System Tumors Located in Difficult to Surgically Access Regions of the Brain and Recurrent/Resistant Pediatric Central Nervous System Tumors Located Anywhere Within the Brain
Brief Title: Laser Interstitial Thermal Therapy (LITT) for the Treatment of Pediatric Central Nervous System Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Anne Bendel, Pediatric Oncologist, Director of Neurooncology, Children's Hospitals and Clinics of Minnesota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1504-044
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser interstitial thermotherapy (LITT) treated patients (Experimental): All patients enrolled on the trial will undergo LITT therapy per protocol. Side-effects and outcomes will be monitored and compared with disease matched historical controls.
  Interventions: Device: Laser Interstitial Thermotherapy (LITT)

INTERVENTIONS:
Device: Laser Interstitial Thermotherapy (LITT) — Magnetic resonance imaging (MRI)-guided laser interstitial thermal therapy (LITT) is a minimally invasive surgical option to treat CNS tumors. LITT uses laser energy delivered to a target (i.e. CNS tumor) through a fiberoptic catheter, which results in damage to intracellular proteins and DNA, and subsequent cell death. LITT provides a sharp demarcation between ablated and unharmed tissue, which, when combined with the ability to monitor and control the ablation via MR thermal imaging, results in a high level of precision and control.
  Other Names: Visualase; Neuroblate

SUMMARY:
Laser Interstitial Thermal Therapy (LITT) is a minimally invasive surgical technique that allows for biopsy and thermal ablation of brain tumors. Pediatric patients with brain tumors who are eligible and enroll in the trial will undergo LITT at the time of diagnosis or at the time of recurrence/progression rather than undergo an open craniotomy and tumor resection/biopsy. LITT will include a stereotactic biopsy followed by thermal ablation of the tumor. This study will monitor the safety and efficacy of LITT for the treatment of pediatric brain tumors.

DETAILED DESCRIPTION:
Pediatric brain tumors have a variety of surgical options depending on the location and type of tumor. Complete or near complete surgical removal of pediatric brain tumors usually results in the best chance of survival or long-term control of the tumor. Surgical resection through an open craniotomy is the most common surgical treatment for accessible brain tumors. For tumors that are not surgically accessible or that are resistant to surgical intervention, treatment is limited to radiation and or chemotherapy, which can have significant long term toxicity in children.

Laser interstitial thermal therapy (LITT) offers a minimally invasive surgical option to treat central nervous system (CNS) tumors. LITT uses laser energy delivered to a target (i.e. CNS tumor) through a fiberoptic catheter, which results in damage to intracellular proteins and DNA, and subsequent cell death. LITT provides a sharp demarcation between ablated and unharmed tissue, which, when combined with the ability to monitor and control the ablation via MR thermal imaging, results in a high level of precision and control. LITT may offer a treatment option for patients with deep brain lesions that are surgically inaccessible, such as tumors located in the thalamus, hypothalamus, basal ganglia and brainstem. LITT may also be a potential treatment for brain tumors which have recurred or persist despite conventional therapies including craniotomy. The MRI-guided laser probe used in LITT utilizes a much smaller surgical corridor through the brain to reach a deep lesion, potentially reducing the risk of complications.

This study will offer LITT, rather than open craniotomy, for the diagnosis and treatment of newly diagnosed pediatric brain tumors located in difficult to surgically access regions of the brain and for the treatment of recurrent/resistant pediatric brain tumors located anywhere within the brain. The primary aim of this study is to determine if LITT is effective in reducing (or at least maintaining current rates of) tumor re-growth while lowering rates of post-surgical complications and improving quality of the procedure (i.e. shorter hospitalization and less use of pain medication compared to standard surgery for tumor removal/biopsy).

This study has the following goals:

1. Determine the frequency of post-operative side-effects in pediatric patients with newly diagnosed, difficult to surgically access CNS tumors or resistant/recurrent CNS tumors in any location who receive LITT treatment for tumor ablation.
2. Examine the role of LITT in controlling newly diagnosed difficult to surgically access CNS tumors or resistant/recurrent pediatric CNS tumors in any location.
3. Assess the correlation between the extent of tumor ablation and the rate of local tumor control.
4. Characterize the MRI changes that occur in a pediatric tumor following LITT ablation.

Patients enrolled on this study will require routine post-LITT follow-up, including intermittent physical exams to assess for side effects and MRIs to monitor the status of the tumor. The follow-up is similar to that performed following an open craniotomy and does not involve any extra studies. The side effects and rate of tumor control for each brain tumor patient enrolled on the trial will be compared to disease matched historical controls to learn more about the morbidity and efficacy of LITT in this population of patients compared to patients who underwent open craniotomy for resection/biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 and 22 years.
2. Karnofsky Performance Scale (for patients > 12 y/o) or Lansky Performance Score (for patients < 12y/o) must be > 50 assessed within two-weeks prior to enrollment.
3. Tumor volume less than 10 cm3 is mandatory for high grade tumors.
4. Tumor volume greater than 10 cm3 is acceptable in low grade tumors if the entire tumor can be ablated in more than one staged procedure.
5. Histology must be available, obtained either at a prior surgery or at the time of LITT by stereotactic biopsy (except in germ cell tumors where elevation of tumor markers is diagnostic).
6. Patients must meet the following histological and disease states:

A) Newly diagnosed low-grade CNS tumor located in a site that is difficult to access surgically or recurrent/persistent low-grade CNS tumor (any site) despite treatment with conventional therapy. Tumor types include:

1. Grade I or II glioma,
2. Desmoplastic neuroectodermal tumor (DNET),
3. Ganglioglioma,
4. Desmoplastic infantile ganglioglioma/astrocytoma,
5. Choroid plexus papilloma (CPP),
6. Meningioma,
7. Subependymal giant cell astrocytoma (SEGA),
8. Craniopharyngioma
9. Teratoma, or
10. Other "low-grade CNS tumors"

B) Newly diagnosed high-grade CNS tumor located in a site that is difficult to access surgically or recurrent/persistent high-grade CNS tumors (any site) despite treatment with conventional therapy. Tumor types include:

1. Grade III or IV glioma,
2. Ependymoma,
3. Atypical teratoid rhabdoid tumor (ATRT),
4. Choroid plexus carcinoma (CPC),
5. Germ cell tumor (GCT),
6. Medulloblastoma/primitive neuroectodermal tumor (PNET),
7. Other "high grade CNS tumors".

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2020-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Morbidity of LITT for the treatment of pediatric brain tumors | 10 years
  The side-effects of LITT for the treatment of pediatric brain tumors will be monitored and compared with disease matched historical controls who underwent open craniotomy for resection or biopsy.
Efficacy of LITT for the treatment of pediatric brain tumors | 10 or more years
  Rates of recurrence or progression of patients treated with LITT for the treatment of pediatric brain tumors will be compared with disease matched historical controls who underwent open craniotomy for resection or biopsy

SECONDARY OUTCOMES:
Tumor control based on extent of tumor ablation | 10 or more years
  Each patient will undergo an MRI thermal map defining the volume of ablated tumor. This volume will be assessed to determine if it is a predictive factor for tumor recurrence or progression.
Characterization of the MRI changes following LITT tumor ablation | 10 years
  The MRI changes that occur following ablation of pediatric brain tumors will be characterized and compared with the MRI findings previously described in adult brain tumors following LITT therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Bendel, M.D., Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States